CLINICAL TRIAL: NCT00565500
Title: A Placebo-Controlled, Double-Blind, Randomized Study of the Potential Interaction Between Aspirin and Ibuprofen or Celecoxib.
Brief Title: Celecoxib, Ibuprofen and the Antiplatelet Effect of Aspirin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Chieti (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Raffaele De Caterina, MD, PhD, G. d'Annunzio University - Chieti
Organization: G. d'Annunzio University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 635-IFL-0508-017; N49-98-71-900
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Ischemic Heart Disease; Osteoarthritis
MeSH Terms: conditions — Myocardial Ischemia; Osteoarthritis | interventions — Celecoxib; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: celecoxib
- 2 (Experimental)
  Interventions: Drug: ibuprofen
- 3 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: celecoxib — celecoxib capsules 200 mg bid for 1 week
  Arms: 1
Drug: ibuprofen — ibuprofen tablets 600 mg tid for 1 week
  Arms: 2
Drug: placebo — placebo capsules tid for 1 week
  Arms: 3

SUMMARY:
Study design: Single center, placebo-controlled, double blind, parallel groups. To evaluate the potential interaction between aspirin and ibuprofen or celecoxib in patients with osteoarthritis (OA) and documented stable ischemic heart disease, a total of 24 patients chronically treated with aspirin will be randomly assigned to one of the 3 treatment groups: 1) celecoxib 200 mg bid; 2) ibuprofen 600 mg tid; 3) placebo.

DETAILED DESCRIPTION:
Patients with arthritis and vascular disease may receive both NSAIDs and lowdose aspirin for the secondary prevention of important vascular events. The use of COX-2 inhibitors may have the potential advantage vs. nonselective NSAIDs in reducing the probability of interfering with permanent inactivation of COX-1 platelet by low-dose aspirin, in this setting. In fact, recent studies suggest that the likelihood of COX-inhibitors to present this pharmacodynamic interaction is inversely related to their COX-2 selectivity. Thus, differently from the non-selective NSAID ibuprofen, prior administration of the selective COX-2 inhibitor rofecoxib, does not antagonize the irreversible inhibition induced by aspirin in healthy subjects. Aim of this study is to determine whether celecoxib given at therapeutic dose at steady state alters the antiplatelet activity of low-dose aspirin, in comparison with ibuprofen.

ELIGIBILITY:
Inclusion Criteria:

1. male or female, age 18-75;
2. subjects with osteoarthritis and documented stable ischemic heart disease;
3. the patient is on long-term aspirin prophylaxis for the ischemic condition;
4. the patient requires or is eligible for chronic treatment with an antiinflammatory and/or analgesic drugs given to control osteoarthritis symptoms;
5. female subjects of childbearing potential must have a negative pregnancy test, use adequate contraception during the study and not be lactating;
6. written informed consent before undergoing any study procedure.

Exclusion Criteria:

1. active gastrointestinal disease (e.g. Crohn's disease or ulcerative colitis) or any evidence of concomitant disease which may lead to early termination of the study;
2. history of active peptic ulceration, gastrointestinal bleeding, esophageal, gastric or duodenal ulcer;
3. known hypersensitivity to COX-2 inhibitors, analgesics, antipyretics, sulfonamides or NSAIDs;
4. treatment with any investigational drug within the previous 30 days;
5. previous participation in this study;
6. evidence of neoplasm or any other severe disease of any organ, including any psychiatric illness;
7. clinically relevant deviations from the normal range in laboratory tests;
8. recent history or suspicion of alcohol abuse or drug addiction;
9. subjects unlikely to be collaborative or to give reliable answers;
10. pregnancy or lactation; female or childbearing potential without a clinical accepted contraceptive method;
11. any severe pathology that can interfere with the treatment or the clinical or instrumental tests of the trial;
12. intake of antiaggregant, anticoagulant, diuretic, beta-blocker, ACE- inhibitor, lithium, methotrexate, cimetidine, digoxin;
13. contraindications to NSAIDs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-04; Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
serum thromboxane (TX)B2 | 1 week

SECONDARY OUTCOMES:
urinary 11-dehydro-thromboxane (TX)B2, arachidonic acid- and ADP-induced platelet aggregation by Born's aggregometer, whole-blood aggregation in the platelet function analyzer (PFA) system, LPS-stimulated prostaglandin(PG)E2 | 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele De Caterina, MD, PhD, Principal Investigator — Institute of Cardiology, G. d'Annunzio University
Locations (1):
- Ce.S.I., Center of Excellence on Aging, G. d'Annunzio University, Chieti, CH, Italy

REFERENCES:
- [Background] Patrono C, Coller B, Dalen JE, FitzGerald GA, Fuster V, Gent M, Hirsh J, Roth G. Platelet-active drugs : the relationships among dose, effectiveness, and side effects. Chest. 2001 Jan;119(1 Suppl):39S-63S. doi: 10.1378/chest.119.1_suppl.39s. No abstract available. PMID 11157642
- [Background] Patrignani P, Filabozzi P, Patrono C. Selective cumulative inhibition of platelet thromboxane production by low-dose aspirin in healthy subjects. J Clin Invest. 1982 Jun;69(6):1366-72. doi: 10.1172/jci110576. PMID 7045161
- [Background] Catella-Lawson F, Reilly MP, Kapoor SC, Cucchiara AJ, DeMarco S, Tournier B, Vyas SN, FitzGerald GA. Cyclooxygenase inhibitors and the antiplatelet effects of aspirin. N Engl J Med. 2001 Dec 20;345(25):1809-17. doi: 10.1056/NEJMoa003199. PMID 11752357
- [Background] FitzGerald GA, Patrono C. The coxibs, selective inhibitors of cyclooxygenase-2. N Engl J Med. 2001 Aug 9;345(6):433-42. doi: 10.1056/NEJM200108093450607. No abstract available. PMID 11496855